CLINICAL TRIAL: NCT01606397
Title: The Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Multiple Escalating Doses of LY2409021 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Multiple Increasing Doses of LY2409021 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11071; I1R-FW-GLBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo administered orally once daily for 4 weeks
  Interventions: Drug: Placebo
- 5 mg LY2409021 (Experimental): 5 mg LY2409021 administered orally once daily for 4 weeks
  Interventions: Drug: LY2409021
- 30 mg LY2409021 (Experimental): 30 mg LY2409021 administered orally once daily for 4 weeks
  Interventions: Drug: LY2409021
- 60 mg LY2409021 (Experimental): 60 mg LY2409021 administered orally once daily for 4 weeks
  Interventions: Drug: LY2409021
- 90 mg LY2409021 (Experimental): 90 mg LY2409021 administered orally once daily for 4 weeks
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: Placebo — Administered orally (capsule)
  Arms: Placebo
Drug: LY2409021 — Administered orally (capsule)
  Arms: 30 mg LY2409021; 5 mg LY2409021; 60 mg LY2409021; 90 mg LY2409021

SUMMARY:
The study drug LY2409021 is being evaluated as a possible treatment for diabetes. The primary purpose of this study is to help answer the following research questions, and not to provide treatment for diabetes :

* The safety of LY2409021 and any side effects that might be associated with it following 4 weeks of doses
* How long it takes the body to absorb and remove LY2409021 following dosing over 4 weeks
* How daily dosing of LY2409021 affects blood levels of sugar (glucose), insulin and other naturally occurring substances before and after a meal
* How LY2409021 works when given with metformin
* How daily dosing of LY2409021 affects the cells that produce insulin

ELIGIBILITY:
Inclusion Criteria:

* Must be either a male, or a female who cannot become pregnant, who has type 2 diabetes and is either controlling diabetes through diet and exercise, or taking metformin
* Have an hemoglobin A1c (HbA1c) value at screening of greater than or equal to 6.5% and less than or equal to 10.0% on a stable treatment regimen at the time of measurement
* Have a screening body mass index (BMI) of 20 to 40 kg/m^2 inclusive
* Have a blood pressure reading at screening of between 90 to 160 millimeters of mercury (mmHg) (systolic) and 40 to 95 mmHg (diastolic)

Exclusion Criteria:

* Have used insulin for diabetic control within 1 year of study entry
* Have used thiazolidinediones within 3 months, or any other drugs for treatment of hyperglycemia (except metformin) within 1 month, prior to first planned dosing. Metformin is acceptable for this study.
* Have clinically significant coronary artery disease
* Have clinically significant peripheral vascular disease
* Have clinical evidence of active diabetic proliferative retinopathy
* Have known significant autonomic neuropathy as evidenced by urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis
* Impaired renal function (serum creatinine greater than 115 micromoles/liter [μmol/L] [1.3 mg/dL] in women, greater than 130 μmol/L [1.5 mg/dL] in men)
* Have triglycerides greater than 4.5 millimoles per liter (mmol/L) [approximately 400 mg/dL] at screening
* Were hospitalized for poor control of diabetes (keto-acidotic episode) in the last 6 months
* Are allergic to LY2409021 or similar drugs
* Have history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (other than diabetes), hematological, or neurological disorders capable of significantly altering the absorption, or metabolism or elimination of drugs or of constituting a risk when taking the study medication or interfering with the interpretation of data
* Have used systemic glucocorticoids within 1 month prior to first dosing
* Have donated 450 mL or more of blood in the last 3 months or have donated any blood within the last month
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female), or are unwilling to stop alcohol as required by the study restrictions (1 unit = 360 mL of beer, or 150 mL of wine, or 45 mL of spirits)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more drug related adverse events (AEs) or any serious AEs | From first dose of study drug up to discharge (at least 28 days after last dose)

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration curve (AUC) of LY2409021 | From first study drug dose to Day 28 post last dose
Pharmacokinetics: Maximum concentration (Cmax) of LY2409021 | From first study drug dose to Day 28 post last dose
Change in fasting blood glucose level | From Day -1 to Day 28 of dosing
Change in incremental area under the curve (AUC) for glucose | From Day -1 to Day 28 of dosing
Change in homeostasis model assessment of beta cell function (HOMA-B) | From baseline to Day 28
Change in fasting glucagon level | From Day -1 to Day 28 of dosing
Change in fasting insulin level | From Day -1 to Day 28 of dosing
Change in fasting C-peptide level | From Day -1 to Day 28 of dosing
Change in fasting glucagon-like peptide-1 (GLP-1) level | From Day -1 to Day 28 of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, United Kingdom

REFERENCES:
- [Derived] Kelly RP, Garhyan P, Raddad E, Fu H, Lim CN, Prince MJ, Pinaire JA, Loh MT, Deeg MA. Short-term administration of the glucagon receptor antagonist LY2409021 lowers blood glucose in healthy people and in those with type 2 diabetes. Diabetes Obes Metab. 2015 Apr;17(4):414-22. doi: 10.1111/dom.12446. Epub 2015 Mar 2. PMID 25656305